CLINICAL TRIAL: NCT02685683
Title: A Phase 2, Open-label Study to Explore the Pharmacodynamic and Clinical Effects of Mongersen (GED-0301) in Subjects With Active Crohn's Disease
Brief Title: Pharmacodynamic and Clinical Outcome Study of Mongersen in Patients With Crohn's Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated by Sponsor following a recommendation from external DMC to terminate the ongoing Phase 3 CD studies; there were no new emergent safety findings
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GED-0301-CD-005
Record Dates: First submitted 2016-02-15; First posted 2016-02-19 (Estimated); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease; GED-0301; Open-label; Pharmacodynamic; Mongersen
MeSH Terms: conditions — Crohn Disease | interventions — GED0301

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GED-0301 Induction (160mg) followed by intermittent 160 mg (Experimental): GED-0301 160 mg "by mouth" (PO) daily (QD) for 12 weeks, followed by alternating GED 0301 160 mg QD for 4 weeks and no IP for 4 week, up to Week 100
  Interventions: Drug: GED-0301

INTERVENTIONS:
Drug: GED-0301 — During Induction period patient will receive mongersen 160 mg daily for 12 weeks. This study also offers subjects the option to continue with maintenance treatment at the discretion of the Investigator, beginning after the Week 12 Visit with alternating no IP for 4 weeks, followed by mongersen (GED-0301) 160 mg QD for 4 weeks, up through the Week 52 Visit during the Maintenance Period. At Week 52, subjects who have achieved an endoscopic improvement of >50% from baseline based on the SES-CD, as assessed by the central reader, and clinical improvement (HBI <7), will have the option to continue receiving treatment for an additional year, up through Year 2 (ie, the Week 100 Visit).
  Other Names: Mongersen

SUMMARY:
This study is designed to explore mechanism of action of mongersen (GED-0301) 160 mg once daily in patients with active Crohn's Disease

DETAILED DESCRIPTION:
Subjects will be screened to provide 20 enrolled subjects who complete 12 weeks of mongersen (GED-0301) 160 mg QD treatment as open-label therapy.

The study will consist of 4 periods:

* Screening Period - up to 4 weeks
* Induction Period - 12 weeks (Week 0 Visit through Week 12 Visit)
* Maintenance Period - 88 weeks (after Week 12 Visit through Week 100 Visit)
* Follow-up Period - 4 weeks (ie, no IP taken)

Subjects who prematurely discontinue treatment from this study prior to Week 100 will have an Early Termination Visit and also enter the 4-week Follow-up Period.

At the Screening Visit, all subjects who meet the entrance criteria will be eligible to enter the study. The number of subjects with previous exposure to Tumor Necrosis Factor-Alpha (TNF-α) blockers is targeted to be approximately 40% (ie, approximately 8 subjects).

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years of age.
* Active Crohn's disease (CD) disease as determined by the Crohn's Disease Activity Index (CDAI) score and the Simple Endoscopic Score for Crohn's Disease (SES-CD)
* Subject must have failed or experienced intolerance to at least one of the following: budesonide; systemic corticosteroids; immunosuppressants (eg, azathiopurine, 6-mercaptopurine, or methotrexate); or biologics for the treatment of CD.
* Subject must use protocol approved contraception

Exclusion Criteria:

* Diagnosis of ulcerative colitis (UC), indeterminate colitis, ischemic colitis, microscopic colitis, radiation colitis or diverticular disease-associated colitis
* Crohn's Disease (CD) manifestations such as abscesses, short bowel syndrome; or intestinal strictures with prestenotic dilatation, requiring procedural intervention or not passable with an adult colonoscope.
* Intestinal resection within 6 months or any intra-abdominal surgery within 3 months prior to the Screening Visit
* Ileostomy or a colostomy
* Prior treatment with more than 2 TNF-α blockers (eg, infliximab or adalimumab).
* Prior treatment with any integrin antagonists (eg, natalizumab or vedolizumab).
* Subject is pregnant or breastfeeding.
* Subject has received prior treatment with mongersen (GED-0301), or participation in a clinical study involving mongersen (GED-0301).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-04-04 (Actual); Primary Completion 2017-09-25 (Actual); Study Completion 2017-11-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline of Smad7 (Mothers Against Decapentaplegic homolog 7) expression in the intestinal mucosa | Baseline and Week 12
  Smad7 is a protein important in cell interactions and stands for "Mothers against decapentaplegic homolog 7" protein

SECONDARY OUTCOMES:
Change from baseline in messenger ribonucleic acid (mRNA) expression of inflammatory cytokines | Baseline and Week 12
  Change from baseline in the mRNA expression of inflammatory cytokines such as, but not limited to, interleukin (IL)-10, IL-25, chemokine (C-C motif) ligand 20 (CCL20) and tumor necrosis factor alpha (TNF-α) in the intestinal mucosa at Week 12, from biopsy samples during ileocolonoscopy
The proportion of subjects achieving clinical remission, defined as a Crohn's Disease Activity Index (CDAI) score < 150, at Weeks 4, 8, and 12 | Up to week 12
  The CDAI is a measure of disease activity in patients with Crohn's Disease.
Change from baseline in the Simple Endoscopic Score for Crohn's Disease (SES-CD) at Week 12 and 52 | Week 12 and week 52
  The SES-CD is a measure that indicates mucosal inflammation in the end part of the ileum (or small intestine) and colon (or large intestine) in patients with Crohn's Disease
Number of Adverse Events | Up to Week 56
  The evaluation of safety and tolerability of GED-0301, assessed by the type, frequency and severity of adverse events, and its relationship to investigational product (IP), discontinuation due to adverse events, and clinically significant changes in electrocardiograms (ECGs), vital signs, and/or laboratory findings

CONTACTS AND LOCATIONS:
Overall Officials: Keith Usiskin, MD, Study Director — Celgene
Locations (2):
- Italy (2):
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Policlinico Tor Vergata, Rome

REFERENCES:
- [Derived] Marafini I, Stolfi C, Troncone E, Lolli E, Onali S, Paoluzi OA, Fantini MC, Biancone L, Calabrese E, Di Grazia A, Monteleone I, Lenti MV, Di Sabatino A, Monteleone G. A Pharmacological Batch of Mongersen that Downregulates Smad7 is Effective as Induction Therapy in Active Crohn's Disease: A Phase II, Open-Label Study. BioDrugs. 2021 May;35(3):325-336. doi: 10.1007/s40259-021-00482-x. Epub 2021 Apr 19. PMID 33871807